CLINICAL TRIAL: NCT01934842
Title: A Study to Compare Analyte Levels in Blood Samples Collected Using the TAP20-C Device With Results Obtained by Fingerstick Using the SAFE-T-FILL Capillary Blood Collection System
Brief Title: A Study to Compare Analyte Levels in Blood Collected Using an Investigational Collection Device With a Commercial Predicate
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Seventh Sense Biosystems (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-P005
Record Dates: First submitted 2013-08-30; First posted 2013-09-04 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes; Anemia
MeSH Terms: conditions — Diabetes Mellitus; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP20-C (Experimental): TAP20-C
  Interventions: Device: TAP20-C
- SAFE-T-FILL (Active Comparator): SAFE-T-FILL
  Interventions: Device: SAFE-T-FILL

INTERVENTIONS:
Device: TAP20-C
  Arms: TAP20-C
Device: SAFE-T-FILL
  Arms: SAFE-T-FILL

SUMMARY:
This study will compare blood collection from the forearm using an investigational device, TAP20-C to blood collection from the finger tip. The blood collected from the forearm and from the fingertip will then be analyzed for glucose, hemoglobin and hemoglobin A1c.

ELIGIBILITY:
Inclusion Criteria:

Healthy Subject Group

1. Male and female volunteers 18 years of age or older.
2. Voluntary written consent to participate in this study.

Diabetic Subject Group

1. Male and female volunteers 18 years of age or older.
2. Have been diagnosed with Type 1 or Type 2 diabetes mellitus by self-report.
3. Voluntary written consent to participate in this study.

Exclusion Criteria:

1. Subjects who are pregnant or nursing mothers by self-report.
2. Subjects who have eaten or consumed sugar-containing drinks in the 2 hours before blood sample collection begins.
3. Subjects with a history of skin disorders or who present with abnormal skin integrity or atypical skin health within the areas to be tested.
4. Subjects with a missing index or middle finger on either hand or a missing forearm
5. Subjects who have known allergies to titanium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Non Inferiority of Analyte Levels | Day 1
  The study will compare the concentrations of glucose, hemoglobin and hemoglobin A1c in blood samples collected with the two different blood collection methods in a single 2 1/2 hour session.

CONTACTS AND LOCATIONS:
Locations (1):
- Seventh Sense Biosytems, Cambridge, Massachusetts, United States